CLINICAL TRIAL: NCT02673593
Title: A Randomised, Double-Blind, Placebo-Controlled, Single Ascending Dose and Multiple Dose Phase I Study to Assess the Safety, Pharmacokinetics and Effect of Food on Orally Administered DS102 in Healthy Subjects
Brief Title: Safety and Efficacy Study of Orally Administered DS102 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DS Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: DS102A-01
Record Dates: First submitted 2016-01-21; First posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Safety; Pharmacokinetics; Food Effect

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Placebo (Placebo Comparator): Taken orally as a single dose (Cohorts 1 - 4) Taken orally as a multiple daily dose for 28 days (Cohorts 5 - 7)
  Interventions: Drug: Placebo
- DS102 100mg Single Dose (Experimental): Taken orally once by Cohort 1
  Interventions: Drug: DS102
- DS102 500mg Single Dose (Experimental): Single Dose taken orally on three separate occasions by Cohort 2 (second and third dose assessing food effect)
  Interventions: Drug: DS102
- DS102 1000mg Single Dose (Experimental): Taken orally once by Cohort 3
  Interventions: Drug: DS102
- DS102 2000mg Single Dose (Experimental): Taken orally once by Cohort 4
  Interventions: Drug: DS102
- DS102 500mg Multiple Dose (Experimental): Taken orally once a day for 28 days by Cohort 5
  Interventions: Drug: DS102
- DS102 1000mg Multiple Dose (Experimental): Taken orally once a day for 28 days by Cohort 6
  Interventions: Drug: DS102
- DS102 2000mg Multiple Dose (Experimental): Taken orally once a day for 28 days by Cohort 7
  Interventions: Drug: DS102

INTERVENTIONS:
Drug: DS102
  Arms: DS102 1000mg Multiple Dose; DS102 1000mg Single Dose; DS102 100mg Single Dose; DS102 2000mg Multiple Dose; DS102 2000mg Single Dose; DS102 500mg Multiple Dose; DS102 500mg Single Dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to investigate the safety, pharmacokinetics and food effect of DS102 (up to 2000mg single and multiple daily doses) and placebo in healthy participants.

DS102 capsules will be orally administered for up to 4 weeks, and will be compared against placebo.

The study will enrol approximately 56 adult subjects.

DETAILED DESCRIPTION:
There will be 7 cohorts enrolled, each consisting of 8 subjects.

Cohorts 1 - 4 will be orally administered up to 2000mg single doses of DS102 on Day 1.

Cohorts 5 - 7 will be orally administered up to 2000mg multiple daily doses of DS102 for 28 days.

The primary objective is to assess the safety and plasma pharmacokinetics of single and multiple daily oral doses of DS102.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and is aged between 18 and 45 years inclusive.
* Subject's body mass index (BMI) is between 18.0 and 30.0 kg/m2 inclusive.
* Subject is a non-smoker, has been a non-smoker for 3 months prior to screening and has a negative urine cotinine test at screening.

Exclusion Criteria:

* Subject has had a clinically significant illness in the 4 weeks before screening.
* Use of prescribed medication in the 2 weeks before dosing or over-the-counter preparations (including vitamins and supplements) for 1 week before dosing
* Subject has a significant history of drug/solvent abuse, or a positive drugs of abuse (DOA) test at screening or Day -1.
* Subject with a history of alcohol abuse in the opinion of the Investigator, or who currently drinks in excess of 28 units per week (males) or 21 units per week (females), whereby a unit consists of 10ml or 8mg of pure alcohol, or who have a positive alcohol urine test at screening or Day -1.
* Subject has participated in any other clinical study with an investigational drug/device within 3 months before the first day of administration of study treatment.
* Subject has a positive test for human immunodeficiency virus (HIV) antibodies, Hepatitis B surface antigen or Hepatitis C antibodies at screening.
* Subject has had a serious adverse reaction or significant hypersensitivity to any drug.
* Subject has donated blood or blood products within 3 months before screening.
* Subject has known hypersensitivity to any ingredients of the study treatment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety (adverse events, laboratory tests, vital signs, ECGs) of DS102 administered as a single dose | 14 days
  Phase I study - Overall safety of product in first in man study
Pharmacokinetics (Plasma concentrations assessed by Cmax) of DS102 administered as a single dose | 14 days
  Phase I study - Overall PK of product in first in man study
Pharmacokinetics (Plasma concentrations assessed by tmax) of DS102 administered as a single dose | 14 days
  Phase I study - Overall PK of product in first in man study
Pharmacokinetics (Plasma concentrations assessed by AUC0-inf) of DS102 administered as a single dose | 14 days
  Phase I study - Overall PK of product in first in man study
Pharmacokinetics (Plasma concentrations assessed by AUClast) of DS102 administered as a single dose | 14 days
  Phase I study - Overall PK of product in first in man study
Pharmacokinetics (Plasma concentrations assessed by CL/F) of DS102 administered as a single dose | 14 days
  Phase I study - Overall PK of product in first in man study
Pharmacokinetics (Plasma concentrations assessed by Vz/F ) of DS102 administered as a single dose | 14 days
  Phase I study - Overall PK of product in first in man study
Pharmacokinetics (Plasma concentrations assessed by t½) of DS102 administered as a single dose | 14 days
  Phase I study - Overall PK of product in first in man study
Safety (adverse events, laboratory tests, vital signs, ECGs) of DS102 administered as a multiple dose for 28 days | 42 days
  Phase I study - Overall safety of product in first in man study
Pharmacokinetics (Plasma concentrations assessed by Cmax) of DS102 administered as a multiple dose | 42 days
  Phase I study - Overall PK of product in first in man study
Pharmacokinetics (Plasma concentrations assessed by tmax) of DS102 administered as a multiple dose | 42 days
  Phase I study - Overall PK of product in first in man study
Pharmacokinetics (Plasma concentrations assessed by AUC0-inf) of DS102 administered as a multiple dose | 42 days
  Phase I study - Overall PK of product in first in man study
Pharmacokinetics (Plasma concentrations assessed by AUClast) of DS102 administered as a multiple dose | 42 days
  Phase I study - Overall PK of product in first in man study
Pharmacokinetics (Plasma concentrations assessed by CL/F) of DS102 administered as a multiple dose | 42 days
  Phase I study - Overall PK of product in first in man study
Pharmacokinetics (Plasma concentrations assessed by Vz/F) of DS102 administered as a multiple dose | 42 days
  Phase I study - Overall PK of product in first in man study
Pharmacokinetics (Plasma concentrations assessed by AUC 0-24) of DS102 administered as a multiple dose | 42 days
  Phase I study - Overall PK of product in first in man study
Pharmacokinetics (Plasma concentrations assessed by Css) of DS102 administered as a multiple dose | 42 days
  Phase I study - Overall PK of product in first in man study
Pharmacokinetics (Plasma concentrations assessed by t½) of DS102 administered as a multiple dose | 42 days
  Phase I study - Overall PK of product in first in man study

CONTACTS AND LOCATIONS:
Locations (1):
- DS Biopharma Investigational Site, Belfast, Ireland